CLINICAL TRIAL: NCT03581656
Title: ChordArt System Study for the Treatment of Mitral Regurgitation Due to Leaflet Prolapse or Flail
Brief Title: ChordArt System for Mitral Regurgitation
Acronym: CHAGALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CoreMedic GmbH (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-000274-001; CHAGALL (Other: Other Identifier)
Record Dates: First submitted 2018-06-04; First posted 2018-07-10 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Mitral Valve Repair; Mitral Regurgitation; Mitral Valve Insufficiency
Keywords: Degenerative Mitral Leaflet Prolapse; Heart Disease; Minimally Invasive
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Single arm, multi-center, prospective, non-randomized study. The study is conducted in accordance with the guidelines of the Mitral Valve Academic Research Consortium (MVARC) regarding study design and endpoint definition as well as International Standards Organization 5840-3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): The ChordArt System is intended for chordal replacement in patients with mitral valve insufficiency due to leaflet prolapse or flail delivered through a catheter based technology for mitral chordal replacement via a small incision in the thorax.
  Interventions: Device: ChordArt System

INTERVENTIONS:
Device: ChordArt System — The ChordArt System is intended for chordal replacement in mitral valve insufficiency due to leaflet prolapse or flail. One or more ChordArt System may be utilized within the same intervention for optimal mitral valve treatment.

SUMMARY:
The ChordArt System is a novel catheter based technology for mitral chordal replacement that enables controlled implantation of artificial mitral chords to treat mitral regurgitation with a minimally invasive approach. The implant is designed to allow transfemoral antegrade implantation.

DETAILED DESCRIPTION:
ChordArt utilizes a minimally invasive catheter based approach by which multiple artificial chordae are precisely positioned into the papillary muscle and then secured to the pathological leaflet.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mitral Regurgitation due to degenerative mitral leaflet prolapse or flail
* Left Ventricular Ejection Fraction >20%
* New York Heart Association functional class II to IV
* Able and willing to give informed consent and follow protocol procedures.

Exclusion Criteria:

* Life expectancy <1 year
* Hemodynamic instability
* Severe untreated ischemic disease
* Pulmonary Hypertension
* Any prior mitral valve surgery or transcatheter mitral valve procedure
* Stroke or transient ischemic event within 30 days before randomization
* Patient is pregnant (urine human chorionic gonadotropin (HCG) test result positive), planning to be pregnant or lactating.
* Renal insufficiency
* Acute anemia
* Chronic obstructive pulmonary disease
* Severe right ventricular dysfunction
* Hepatic insufficiency
* Patient is participating in other investigational studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At 30 days from implant procedure
  The frequency of all-cause mortality
Major adverse events | At 30 days from implant procedure
  The frequency of pre-determined major adverse events

SECONDARY OUTCOMES:
Technical Success | End of Implantation Procedure
  The technical success will be measured by the absence of procedural mortality, successful access, delivery of the ChordArt implant & retrieval of the ChordArt delivery system as well as successful ChordArt deployment, positioning and freedom from emergency surgery or re-intervention related to the device or access procedure.
Device Performance | At 30 days
  The device performance will be measured by the reduction of Mitral Regurgitation by Echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Kestutis Rucinskas, MD, Principal Investigator — Heart Surgery Centre, Santariskiu Vilnius
Locations (1):
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohty D, Orszulak TA, Schaff HV, Avierinos JF, Tajik JA, Enriquez-Sarano M. Very long-term survival and durability of mitral valve repair for mitral valve prolapse. Circulation. 2001 Sep 18;104(12 Suppl 1):I1-I7. doi: 10.1161/hc37t1.094903. PMID 11568020
- [Background] Urbanski PP. Modified technique of chordal replacement for mitral valve repair. Thorac Cardiovasc Surg. 2005 Oct;53(5):315-7. doi: 10.1055/s-2005-865685. PMID 16208620
- See also: Sponsor's Website — http://www.coremedic.ch/about-us/
- See also: Collaborator's Website — https://www.meditrialeurope.com/